CLINICAL TRIAL: NCT01332890
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between Revaprazan and Itopride HCl in Healthy Male Subjects
Brief Title: Pharmacokinetic Drug Interaction Between Revaprazan and Itopride HCl in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YCD192
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Drug interaction; revaprazan; Itopride HCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental)
  Interventions: Other: Sequence 1
- Sequence 2 (Experimental)
  Interventions: Other: Sequence 2
- Sequence 3 (Experimental)
  Interventions: Other: Sequence 3
- Sequence 4 (Experimental)
  Interventions: Other: Sequence 4
- Sequence 5 (Experimental)
  Interventions: Other: Sequence 5
- Sequence 6 (Experimental)
  Interventions: Other: Sequence 6

INTERVENTIONS:
Other: Sequence 1 — Period1(A) Period2(B) Period3(C) A : Revaprazan 200mg/Day (multiple dose for 7days) B : Itopride 50mg/Day (multiple dose for 7days) C : Revaprazan 200mg plus Itopride 50mg(multiple dose for 7days)
  Arms: Sequence 1
Other: Sequence 2 — Period1(C) Period2(A) Period3(B) A : Revaprazan 200mg/Day (multiple dose for 7days) B : Itopride 50mg/Day (multiple dose for 7days) C : Revaprazan 200mg plus Itopride 50mg(multiple dose for 7days)
  Arms: Sequence 2
Other: Sequence 3 — Period1(B) Period2(C) Period3(A) A : Revaprazan 200mg/Day (multiple dose for 7days) B : Itopride 50mg/Day (multiple dose for 7days) C : Revaprazan 200mg plus Itopride 50mg(multiple dose for 7days)
  Arms: Sequence 3
Other: Sequence 4 — Period1(C) Period2(B) Period3(A) A : Revaprazan 200mg/Day (multiple dose for 7days) B : Itopride 50mg/Day (multiple dose for 7days) C : Revaprazan 200mg plus Itopride 50mg(multiple dose for 7days)
  Arms: Sequence 4
Other: Sequence 5 — Period1(B) Period2(A) Period3(C) A : Revaprazan 200mg/Day (multiple dose for 7days) B : Itopride 50mg/Day (multiple dose for 7days) C : Revaprazan 200mg plus Itopride 50mg(multiple dose for 7days)
  Arms: Sequence 5
Other: Sequence 6 — Period1(A) Period2(C) Period3(B) A : Revaprazan 200mg/Day (multiple dose for 7days) B : Itopride 50mg/Day (multiple dose for 7days) C : Revaprazan 200mg plus Itopride 50mg(multiple dose for 7days)
  Arms: Sequence 6

SUMMARY:
To evaluate drug-drug interaction

DETAILED DESCRIPTION:
The main objective is to evaluate the pharmacokinetic profile of the 50mg Revaprazan plus 50mg Itopride compared to 50mg Revaprazan or 50mg Itopride alone in healthy Korean subjects

ELIGIBILITY:
Inclusion Criteria:

* Males aged 20 to 50 years old, with a body mass index (BMI) between 19 and 27 kg/m2
* Acceptable medical history, physical exam,laboratory tests and EKG, during screening
* Eligible for blood sampling during study period
* Provision of signed written informed consent

Exclusion Criteria:

* History of any clinically significant disease
* History of drug/chemical/alcohol abuse
* Clinically significant illness or within 30days before the first dose
* Use of medication known to chronically alter drug absorption or elimination processes within 30days before the first dose of investigational product
* Use of prescribed medication during the 14 days before administration of the first dose of investigational product
* Use of any non-prescribed medication during the 7 days before administration of the first dose of investigational product - Use of any oriental medication medication during the 30 days before administration of the first dose of investigational product
* Participated in a clinical study involving administration of an investigational drug (new chemical entity) or a marketed drug within past 90 days
* Consuming more than 21 units of alcohol per week
* Smoking more than 20 cigarettes per day or consuming more than 5 cups of caffeinated beverages.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Blood sampling will be obtained on day 7 at each period.
  Serum for each treatment period Experimental. AUCtau, Cmax will be estimated using non-compartmental analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- ASAN Medical Center, University of Ulsan, Seoul, South Korea